CLINICAL TRIAL: NCT03557905
Title: Ultrasonographic Assessment of Lung Recruitment Maneuvers in Pediatric Patients Undergoing Lengthy Microsurgery Operations
Brief Title: Ultrasonographic Assessment of Lung Recruitment Maneuvers in Children Undergoing Lengthy Microsurgery Operations
Acronym: RM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Professor of anesthesia and intensive care, faculty of medicine, Assiut university., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17200202
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Intraoperative Complications
MeSH Terms: conditions — Intraoperative Complications

STUDY DESIGN:
Intervention Model Description: To explore the clinical value of ultrasonic monitoring in the diagnosis of anesthesia-induced atelectasis, the assessment of the effects of lung recruitment, the best positive end-expiratory pressure (PEEP) after RM and in the detection of the point of lung re-collapse after RM in pediatric patients undergoing lengthy microsurgery operations using two levels of intraoperative FIO2 (0.5 VERSUS 0.3).
Who Masked: Participant, Outcomes Assessor
Masking Description: Ventilator adjustments, lung recruitment, PEEP titration and ultrasonographic assessments will be done by well-trained investigators not involved in data collection. The surgeon, the parents or legal guardians and the data collection personell will be blinded to the patients' group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Patients will receive recruitment maneuver (RM) followed by decremental PEEP titration 1min. after establishment of mechanical ventilation and after documented lung re-collapse at an FiO2 of 0.5. .
  Interventions: Device: RM 0.5
- Group II (Active Comparator): Patients will receive recruitment maneuver (RM) followed by decremental PEEP titration 1min. after establishment of mechanical ventilation and after documented lung re-collapse at an FiO2 of 0.3.
  Interventions: Device: RM 0.3

INTERVENTIONS:
Device: RM 0.5 — Patients will receive recruitment maneuver (RM) followed by decremental PEEP titration 1min. after establishment of mechanical ventilation and after documented lung re-collapse.
  Other Names: RM
  Arms: Group I
Device: RM 0.3 — The patient will be ventilated with volume control mode with tidal volume 6 ml/kg, PEEP 3 cmH2O, an inspiratory expiratory ratio of 1:1.5, respiratory rate 20-25 breaths per minute depending on the patient's age and FiO2 of 0.3.
  Other Names: RM
  Arms: Group II

SUMMARY:
The aim of this study will be to explore the clinical value of ultrasonic monitoring in the diagnosis of anesthesia-induced atelectasis, the assessment of the effects of lung recruitment, the best positive end-expiratory pressure (PEEP) after RM and in the detection of the point of lung re-collapse after RM in pediatric patients undergoing lengthy microsurgery operations using two levels of intraoperative FIO2 (0.5 VERSUS 0.3).

DETAILED DESCRIPTION:
* To maximize the benefits, minimize the drawbacks and assess the adequacy of the recruitment maneuver; adequate monitoring at the bedside is essential. Several methods have been proposed, including measuring end-expiratory lung volume or pulmonary compliance, volumetric capnography, oxygenation indices, electrical impedance tomography, computerized tomography and lung ultrasound.
* For lung CT examination patients must be transported out to the radiation unit, which carries risk of transfer, high cost, and radiation exposure. The oxygenation method which is the most commonly used, but it is necessary to repeat arterial blood collection many times, which is cumbersome and expensive.
* Using lung ultrasound (LUS) as real-time guidance during the recruitment maneuver has gained popularity recently owing to its' easy applicability and non-invasive nature. Sonography is a radiation-free methodology which plays an important role in diagnosing pulmonary diseases in children, including obstructive and compressive atelectasis of different origins. Furthermore, lung ultrasound has shown reliable sensitivity and specificity for the diagnosis of anaesthesia-induced atelectasis in children.
* LUS can identify children needing a recruitment maneuver to re-expand their lungs and help optimize ventilator treatment during anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2-12 years old.
* ASA physical status classification I-II.
* Undergoing lengthy microsurgery operations
* and requiring endotracheal intubation and mechanical ventilation for more than 4 hours.-

Exclusion Criteria:

* ASA Physical status classification >II.

  * Thoracic or abdominal surgery.
  * Preexisting lung disease.
  * Pre-operative chest infection or abnormal chest US findings.
  * Cardiac patients.-

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Lung Areation Score | 10 minutes after induction of anesthesia
  lung Areation Score calculated on first lung ultrasound.For a given thoracic area, points will be allocated to the worst LUS pattern observed and video clips of each region examined will be stored. The sum of the points obtained in all the 12 lung areas will define the LUS aeration score, ranging from 0 to 36 for the whole thorax. This score is inversely proportional to the degree of lung aeration.

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdelghaffar, MD, Principal Investigator — Professor of anesthesia, faculty of medicine, Assiut university, Egypt.
Locations (1):
- Assiut university main hospital, Microsurgery unit, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No